CLINICAL TRIAL: NCT06535568
Title: International, Multicenter, Investigator-driven Randomized Clinical Trial to Assess the Single vs. Dual Antiplatelet Therapy in Elderly or HBR Patients Undergoing Percutaneous Intervention With Drug-coated Balloons (PICCOLETO IV-EPIC 38)
Brief Title: Single vs. Dual Antiplatelet Therapy in Elderly or HBR Patients Undergoing Percutaneous Intervention With DCB (PICCOLETO IV-EPIC 38)
Acronym: PIV-EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Ricerca e Innovazione Cardiovascolare ETS (Other)
Collaborators: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICCOLETO IV-EPIC 38
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coronary Disease; Heart Diseases; Cardiovascular Diseases; Myocardial Ischemia; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease; Acute Coronary Syndrome; Coronary Stenosis; Molecular Mechanisms of Pharmacological Action; Enzyme Inhibitors; MTOR Inhibitors; Protein Kinase Inhibitors; Physiological Effects of Drugs; Immunosuppressive Agents; Antineoplastic Agents; High Bleeding Risk; Single Antiplatelet Therapy; Dual Antiplatelet Therapy; Cyclooxygenase Inhibitors; P2Y12 Inhibitor; Platelet Aggregation Inhibitors; Aspirin; Clopidogrel
Keywords: DCB; Angioplasty; Paclitaxel; Antiplatelet treatment; Single antiplatelet therapy (SAPT); Dual antiplatelet therapy (DAPT); High bleeding risk (HBR); MACE; Native CAD; stable or unstable coronary syndromes
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases; Myocardial Ischemia; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease; Acute Coronary Syndrome; Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single antiplatelet therapy (Experimental)
  Interventions: Device: Drug-coated balloon; Drug: Single antiplatelet therapy (SAPT)
- Dual antiplatelet therapy (Active Comparator)
  Interventions: Device: Drug-coated balloon; Drug: Dual antiplatelet therapy (DAPT)

INTERVENTIONS:
Device: Drug-coated balloon — Essential Pro paclitaxel eluting coronary balloon dilatation catheter is a rapid exchange catheter, also known as RX because it has a proximal simple lumen configuration and a distal coaxial dual lumen, intended for coronary arteries percutaneous transluminal angioplasties. Patients assigned to this Arm will be treated with a Drug-Coated Balloon (DCB) after pre-dilatation, the angiography will be conducted as standard of care.
Drug: Single antiplatelet therapy (SAPT) — The antithrombotic regimen is single antiplatelet therapy (SAPT). The Investigator will decide if to use aspirin or clopidogrel, whereas ticagrelor or prasugrel are not recommended in our study population since no benefit (or even harm) has been shown by these drugs in head-to-head trials versus clopidogrel in elderly PCI populations. The type of agent and treatment duration will be selected according to the clinical characteristics of the patient.
  Arms: Single antiplatelet therapy
Drug: Dual antiplatelet therapy (DAPT) — The antithrombotic regimen will follow the standard of care with a dual antiplatelet regimen (DAPT) per local preferences and international guidelines/ARC consensus paper. The type of agent and treatment duration will be selected according to the patient's clinical characteristics.
  Arms: Dual antiplatelet therapy

SUMMARY:
This international, multicenter, open-label, randomized clinical trial evaluates the safety and efficacy of single antiplatelet therapy (SAPT) compared to dual antiplatelet therapy (DAPT) in elderly or high bleeding risk patients undergoing percutaneous coronary intervention (PCI) with the latest generation drug-coated balloon (DCB). The study includes patients with stable or unstable coronary syndromes and aims to assess rates of ischemic and bleeding adverse events.

DETAILED DESCRIPTION:
The purpose of the PICCOLETO IV-EPIC 38 study is to observe and evaluate the efficacy and safety of single antiplatelet therapy (SAPT) after successful PCI with the Essential Pro drug-coated balloon in native coronary artery disease in vessels with a diameter between 2.0 and 4.0 mm, compared to routine dual antiplatelet therapy (DAPT). Patients aged 75 years or older, or those at high bleeding risk, with stable or unstable coronary syndromes will be enrolled and randomized in this study.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients who meet the following criteria:

* Age ≥ 75 years or age ≥ 18 years at high bleeding risk;
* Successful PCI with Essential Pro DCB just performed, in 1, 2 or 3 coronary vessels;
* Stable or unstable coronary syndromes;
* De novo coronary lesions in vessels with diameter ≥2.0 and ≤4.0 mm (visual estimation);
* Informed consent to participate in the study given by the patient or impartial witness.

Exclusion Criteria:

* Stent implantation during index or recent (<6 months) procedure;
* Known (and untreatable) hypersensitivity or contraindication to aspirin, heparin, clopidogrel, paclitaxel or contrast media, or any of their excipient which cannot be adequately pre-medicated;
* Pregnancy at the time of hospitalization;
* Patients participating in another clinical study in which an investigational drug or device was administered within 30 days of screening or within the 5 half-lives of the study drug, whichever is longer;
* ST-elevation myocardial infarction;
* Life expectancy <12 months;
* Left ventricular ejection fraction <30%;
* Visible thrombus at lesion site;
* Target lesion/vessel with any of the following characteristics:

  * severe and/or >270° calcification of the target vessel, also proximal to the lesion (intravascular imaging not mandatory);
  * left main stem stenosis >50%;
  * target lesion is in the left main stem;
  * chronic total occlusion with anticipated necessity of retrograde approach;
  * lesion is in a bypass graft.
* History of asthma induced by the administration of salicylates or substances with a similar action, notably non-steroidal anti-inflammatory medicines (NSAIDs);
* History of gastrointestinal perforation, ulceration, or bleeding (peptic ulcer bleeding-PUBs) related to previous use of NSAIDs or anticoagulant medications, or intracranial hemorrhage;
* Acute gastrointestinal ulcers;
* Hemorrhagic diathesis (including known bleeding disorders or ongoing active bleeding);
* Severe renal impairment (eGFR < 30 mL/min);
* Severe hepatic impairment (Child-Pugh C), with elevated liver enzymes (ALT/AST > 2 x ULN or total bilirubin >1.5 x ULN);
* Severe cardiac failure (NYHA grade III or IV);
* Combination with methotrexate at doses of 15 mg/week or more;
* Patients with baseline neutrophil counts < 1500 cells/mm³;
* Breastfeeding women;
* Full-blown thyrotoxicosis;
* Patients with a very high risk of thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Net Adverse Clinical Events (NACE) at 12 months | 12 months
  Superiority of single antiplatelet therapy (SAPT) versus dual antiplatelet therapy (DAPT) in elderly or high bleeding risk patients undergoing percutaneous coronary intervention (PCI) with drug-coated balloons (DCB), assessed by the rate of Net Adverse Clinical Events (NACE). NACE is defined as the composite of major adverse cardiovascular events (MACE) plus clinically relevant bleeding events classified as BARC 2, 3, or 5, evaluated at 12 months following successful PCI with DCB.

SECONDARY OUTCOMES:
Rate of Clinically Relevant Bleeding Events (Bleeding Academic Research Consortium [BARC] Scale, Grades 2-5; range 0-5, where higher grades indicate more severe bleeding and worse clinical outcome) | 12 months
  Incidence of clinically relevant bleeding events classified as BARC grades 2, 3, or 5 according to the Bleeding Academic Research Consortium (BARC) bleeding definition (scale range 0-5; higher scores indicate worse outcome) in elderly or high bleeding risk patients treated with single antiplatelet therapy (SAPT) versus dual antiplatelet therapy (DAPT) following percutaneous coronary intervention (PCI) with drug-coated balloon (DCB).
Procedural success rate immediately post-PCI | Post-PCI
  Defined as final stenosis <30%, distal TIMI 3 flow, and no major in-hospital adverse events.
Patient-oriented composite endpoint (PoCE) | 12 months
  Composite of all-cause death, all myocardial infarctions (MIs), or any repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Auxologico Milano, Milan, MI, Italy